CLINICAL TRIAL: NCT03271190
Title: Impact of a Cognitive Intervention Enriched With Leisure Activities on Cognition, Daily Life Functioning and Brain Structure and Function in Persons With Subjective Cognitive Decline: The ENGAGE Program
Brief Title: Impact of a Cognitive Intervention Enriched With Leisure Activities in Persons With Subjective Cognitive Decline
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Rotman Research Institute at Baycrest (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Sylvie Belleville, Ph.D, Full professor, University of Montreal, and Scientific Director, Institut Universitaire de Geriatrie de Montreal (IUGM), Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRIUGM-004
Record Dates: First submitted 2016-12-15; First posted 2017-09-05 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Subjective Cognitive Decline
Keywords: aging; memory complaint

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENGAGE SPANISH/MUSIC (Experimental): Cognitive strategies to improve attention and memory skills and application in selected leisure activities (music or Spanish lessons, and videogames) over 4 months.
  Interventions: Behavioral: ENGAGE SPANISH/MUSIC
- ENGAGE DISCOVERY (Active Comparator): Educational program about brain and healthy aging complemented by learning of new information with videogames, documentaries and group discussions over 4 months.
  Interventions: Behavioral: ENGAGE DISCOVERY

INTERVENTIONS:
Behavioral: ENGAGE SPANISH/MUSIC — Cognitive strategies to improve attention and memory skills (21 hours), leisure activities (music lessons or Spanish lessons) (27 hours), selected videogames to practice variable attention strategies (4 hours in class + about 10 hours at home). Total of 24 2-hour in class sessions over 4 months. The training will be delivered to small groups of 5 to 8 participants by a trained therapist for formal sessions and a professional music or Spanish teacher for leisure sessions.
  Arms: ENGAGE SPANISH/MUSIC
Behavioral: ENGAGE DISCOVERY — Educational content about brain and healthy aging (21 hours), leisure activities (watching documentaries followed by group discussion and debate) (27 hours), selected non-stimulating videogames (4 hours in class + about 10 hours at home). Total of 24 2-hour in class sessions over 4 months. The training will be delivered to small groups of 5 to 8 participants by the same trained therapist as in the ENGAGE arm.
  Arms: ENGAGE DISCOVERY

SUMMARY:
The team "Cognitive intervention, cognitive reserve and brain plasticity", Team 10, is part of the Canadian Consortium on Neurodegeneration in Aging (CCNA). The team's aim is to develop and test a multi-faceted intervention program meant to increase cognitive and brain reserve by providing cognitive stimulation through participation in cognitive training sessions and engaging leisure activities. This will be done with a partially randomized controlled double-blind preference trial with a comprehensive cohort design, in participants with subjective cognitive decline (SCD) recruited in Montreal and Toronto.

DETAILED DESCRIPTION:
In the absence of a cure for Alzheimer's disease (AD), there is paramount interest for non-pharmacological cognitive interventions that are designed to restore, increase, or optimize capacities and adaptation. Numerous epidemiological studies have shown that education, cognitively engaging leisure activities, and cognitively demanding professions are associated with a lower risk of cognitive decline and dementia. When estimating the proportion of AD cases attributable to modifiable risk factors, it was found that cognitive inactivity was the factor that contributed to many of the cases worldwide (19.1% or 6.5 million cases). Thus, the level of cognitive stimulation that individuals receive throughout their life is a critical protective factor against cognitive decline and AD, which suggests potentially powerful avenues for intervention. In a number of influential papers, Stern suggested that differences in cognitive lifestyle contribute to cognitive reserve, defined as the built-up resilience of the brain against the detrimental effect of age-related brain damage. Cognitive stimulation is thought to create richer brain networks and facilitate the recruitment of alternative regions or networks. Barnes and Yaffe projected that 1.375 million AD cases worldwide might be prevented by reducing by 25% the prevalence of cognitive inactivity. These findings have tremendous consequences when designing strategies against dementia. Thus, the goal of Team 10 is to design and test an innovative cognitive training program to increase cognitive reserve and reduce decline in persons with a high risk of AD.

Many studies have shown that cognitive training can increase cognitive abilities in healthy older adults, or persons with mild cognitive impairment (MCI). Studies with MCI also show that cognitive training in MCI results in greater brain activation and connectivity, as well as the recruitment of alternative networks, which supports the view that it contributes to the creation of cognitive reserve.

There are different types of cognitive interventions that are potentially available. Choosing the proper one necessitates a fine understanding of their mechanisms of action and their match to the individual's needs and capabilities. Furthermore, many of the existing programs have not received empirical support from studies relying on good quality methodology and there is a lack of evidence regarding their capacity to reduce cognitive decline and dementia. Hence, previous studies have been limited by some or all of the following methodological issues: 1) they most often relied on a small number of participants; 2) they had time-limited follow-up; 3) many did not use a randomized controlled design or provided limited information on their randomization process; 4) very few have assessed the participant characteristics that define best responders (i.e., the profile of individuals that benefit the most from the intervention). Another important aspect is that the programs that are typically used in those studies are often not optimally adapted to seniors' needs and preferences and are not grounded in real life, limiting adherence and generalization to everyday life. Emotional and cognitive engagement refers to participants enjoying as well as actively participating to the learning experience and has been shown to be a critical factor in determining learning outcomes. Thus, our program will be designed to promote engagement, which is absent in the previous studies. Finally, one other important gap is that there are still a lot that is unknown about the brain processes involved in these interventions and how they alter brain structure and/or function, especially in healthy older adults. Thus, an additional important issue is to understand the brain plasticity processes resulting from cognitive training. Brain plasticity refers to the remarkable ability of the central nervous system to spontaneously re-organize or expand during normal learning processes, or to self-repair in acute or progressive brain diseases. This is critical given that an increasing number of studies has revealed that non-pharmacological interventions can have a positive impact in AD and that intermediate mechanisms of neural plasticity and functional compensation likely modulate the detrimental effect of the disease on symptoms.

The investigators will develop ENGAGE, a program to increase cognitive reserve and reduce decline over a 2-year period in persons with a high risk of AD. The investigators propose a multi-faceted intervention program meant to increase reserve by providing cognitive stimulation through participation in engaging cognitive and leisure activities. This ground-breaking program proposes for the first time to combine (1) hands-on training to improve memory and attention through teaching strategies to optimize efficiency, and (2) selected engaging leisure activities that are known to increase brain functions in younger and older adults, such as learning music, learning a second language, and playing carefully selected casual video-games. There are many reasons to combine brain training and leisure activities. First, one limitation of brain training for memory and attention is that participants sometimes fail to generalize the strategies learned in a lab setting and to apply them in their everyday life. Thus, the investigators propose to practice these strategies in the leisure activities, e.g., to learn information relevant to the music or Spanish lessons. Providing natural, ecologically-valid situations to apply and practice the cognitive strategies is done to train participants to use them more spontaneously outside the formal brain training setting. Second, these leisure activities correspond to the cognitively demanding activities that are identified as protective in epidemiological studies, and thus likely to promote brain plasticity. Third, they are attractive and will therefore improve motivation for training. The enjoyable characteristic of the leisure activities will also make them attractive to older adults with lower education, a segment of population which may especially benefit from such intervention. Finally, if proven effective, the training program will have the important advantage of being easy to implement in the community and will be relatively low-cost relative to formal health care. Another objective of this research project is to provide recommendations regarding profiles of participants which may benefit the most from the intervention. The investigators will thus measure whether the effect of the training is modulated by sex differences as women have been suggested to have less brain reserve than men as well as age, education or socio-cultural background, lifestyle habits, genetic factors and other markers of cognitive reserve.

The research team benefits from the contribution of clinicians and researchers from across Canada who will combine their unique expertise on brain training and on the effects of leisure activities on the brain to provide the most innovative and potentially meaningful approach to cognitive intervention. Overall, this innovative program will provide brain training through specific cognitive training and carefully selected leisure activities that are known to have a positive impact on cognition and will be particularly attractive to older adults from varied backgrounds.

Objectives

* Develop a multi-faceted intervention program that combines brain-based cognitive training and engaging leisure activities to increase cognitive reserve.
* Examine whether the program improves cognition and well-being, and prevents cognitive decline.
* Assess its effect on brain structure and function using structural and functional Magnetic Resonance Imaging (fMRI).
* Determine if individual differences (demographics, reserve level, genetic background) modulate outcomes.
* Provide empirical evidence that cognitively-engaging activities provided later in life can increase brain reserve, promote cognitive health and reduce cognitive decline.

Hypotheses. The investigators hypothesize that participants who will be engaged in the intervention program will show better behavioral and brain outcomes than participants from the control group who will receive an active control program. More specifically, improved behavioral performance following the intervention is expected in neuropsychological tests measuring cognitive components that are targeted in the program (mainly memory and attention), as well as a transfer effects to an ecologically-valid test measuring functioning in a simulated real-life situation. The investigators also expect improvement in participants' subjective evaluation of their proficiency and satisfaction with life (questionnaires). Regarding retention of training benefits, the hypothesis is that the experimental group will show better cognition at the follow up testing, 2 years from the beginning of the study, and less cognitive decline when comparing 0- to 2-year performance. Regarding fMRI testing, the investigators expect more task-related activation following training and correlations between brain changes and cognitive gain, which would be considered as a marker of enhanced neurocompensation processes.

Design. The consort guidelines will be used to organize and report the trial (http://www.consort-statement.org). The study uses a randomized controlled double-blind preference trial with a comprehensive cohort design. Outcomes will be tested by assessors who will not be involved in the intervention, and who will be blind to training assignment. One hundred forty-four (144) participants with subjective cognitive decline (SCD), but no objective impairment based on cognitive tests, will be recruited and randomly assigned to either the cognitive program (ENGAGE SPANISH or ENGAGE MUSIC) or the active control program (ENGAGE DISCOVERY). Participants in the ENGAGE DISCOVERY program will undergo the same amount of activities as proposed in the ENGAGE SPANISH/MUSIC programs, but those activities will be designed not to be cognitively challenging. Behavioral measures (objective and subjective measures of cognition and efficiency in everyday life functioning) as well as neuroimaging measures (fMRI scan during a memory task) will be collected at 3 time points: before the intervention (PRE), immediately after the intervention (POST-1), and 2 years after PRE (POST-2). PRE tests will be administered within a 12-week window before the beginning of the intervention. POST-1 and POST-2 will each be administered within a 8-week window.

To ensure that participants will not be enrolled in an activity that they dislike, and thus remain the 'leisure' aspect, they will be able to exclude either the 'Music' or 'Spanish' activity prior to randomization to the intervention or control conditions. This was decided to personalize the intervention as people vary considerably in how attracted they are by different leisure activities, and to give participants a sense of choice, which was found to reduce disappointment related to randomization, and thus to reduce attrition. This will be done in a manner that will allow preserving double blindness. If participants who are randomized in the cognitive program did not wish to exclude an activity, then a second randomization will assign them in one of the 2 activities (either music or Spanish). Thus, the training vs active control comparison is fully randomized but further comparison of the two leisure activities will rely on a partially randomized comparison cohort. In that case, the randomized cohorts will be first compared, followed by a comparison of the entire cohort, including those in the preference arm.

The results of this intervention will be analyzed at three-endpoints: 1) at baseline (PRE); 2) immediately after the intervention (POST-1); and 3) 2 years after baseline, i.e., about 18 months after the end of the intervention (POST-2).

ELIGIBILITY:
Inclusion Criteria:

* Possess sufficient visual and auditory acuity to undergo neuropsychological tests and to do the intervention.
* Commit for the whole intervention + 2 follow-up sessions 2 years from pre-test.
* Have an internet connection at home.
* Answer 'Yes' to both following questions: "Do you feel like your memory is becoming worse?" "Does this worry you?"
* Have a delayed recall score above the education-adjusted cut-offs (≥9 for 16+ years of education; ≥5 for 8-15 years of education; ≥3 for 0-7 years of education) at the Logical Memory test (Wechsler Memory Scale, maximum score 25).
* Have a Montreal Cognitive Assessment (MoCA) total score of 20 and above (≥20/30).
* Have a delayed recall score at the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List task above 4 (>4).
* Have a global Clinical Dementia Rating score (CDR) equal to 0 or 0.5 (=0 to 0.5).

Exclusion Criteria:

* The presence of disease or injury of the central nervous system, such as: moderate to severe chronic static leukoencephalopathy (including previous traumatic injury), multiple sclerosis, a serious developmental handicap, subdural hematoma (past or current), subarachnoid haemorrhage (past or current), primary cerebral tumour or cerebral metastases, epilepsy (current), dementia or another neurodegenerative disease, and other rarer brain illnesses.
* Symptomatic stroke within the previous year.
* History of intracranial surgery.
* Major surgery within last 2 months.
* Serious comorbid condition that, in the opinion of the study investigator, is likely to result in death within a year.
* Major depression or anxiety.
* Schizophrenia or other major psychiatric disorder.
* Ongoing alcohol or drug abuse that in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.
* Subject does not have a study partner who can provide corroborative information.
* Individuals where English (Toronto) or French (Montreal) is not sufficiently proficient for clinical assessment and neuropsychological testing.
* Unable to undergo MRI scan due to medical contraindications or inability to tolerate the procedure.
* Plans on moving outside the province within the next 2 years.
* Musicianship: more than 5 years of formal music training in total life or more than 10 years of choir experience.
* Fluency in Spanish: has learned Spanish after secondary school for more than 5 years, speaks Spanish at home, has ever lived in a Hispanic country.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in episodic memory (composite score) | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  A composite score will be computed by averaging z-scores from the delayed recall of the Rey Auditory Verbal Learning Test (RAVLT) and the delayed recall of the face-name association task (an associative memory test adapted from Simona Brambati's task for the Consortium pour l'Identification precoce de la Maladie d'Alzheimer (CIMA-Q) study currently running in Quebec).

SECONDARY OUTCOMES:
Changes in attention control (composite score) | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  A composite score will be computed by averaging the z-scores from the Number-letter task (switching cost), the complex (4-choice) reaction time from the Canadian Longitudinal Study on Aging (CLSA) Reaction Time Task, and an adapted Flanker task comprising a dual-task condition (congruency effect and dual task cost).
Changes in psychological health: Anxiety and depression (composite score) | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  A composite score will be computed by averaging the z-scores from the Geriatric Anxiety Inventory (GAI) + Geriatric Depression Scale (GDS).
Changes in psychological health: Apathy | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  A composite score will be computed that averaging the z-scores from the participant + informant versions of the Apathy Inventory Scale.
Changes in psychological health: Quality of life (composite score) | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  A composite score will be computed by averaging the z-scores from the 36-item Short Form Survey (SF-36), assessing activities and well-being, and the Quality of Life Alzheimer's Disease questionnaire (QoL-AD).
Changes in psychological health: Help-seeking behaviour | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  Mean scores from the medical care section from the Stanford Chronic Disease questionnaire, related to medical help-seeking behavior.
Changes in brain structure: Hippocampal Volume (for a subgroup of participants) | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  Participants will be scanned on a Siemens Total Imaging Matrix (TIM) Trio 3 T magnetic resonance imaging (MRI) system (Siemens Medical Solutions, Erlangen, Germany). Hippocampal volume (mm3) will be measured, as this is an early biomarker of AD and is found to be a sensitive marker of memory training.
Changes in brain structure: Cortical Thickness (for a subgroup of participants) | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  Participants will be scanned on a Siemens TIM Trio 3 T magnetic resonance imaging (MRI) system (Siemens Medical Solutions, Erlangen, Germany). Cortical thickness (mm) will be measured, as this is an early biomarker of AD and is found to be a sensitive marker of memory training.
Changes in brain function: Brain activation (for a subgroup of participants) | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention)
  fMRI activity while participants are doing an associative memory task. Participants will be presented a sequence of 80 images (e.g., animals, vegetables, etc.). They appear within one of the four quadrants of the screen. People are asked to remember the images and their position among the 4 quadrants (either top-left, top right, bottom-left or bottom-right). Retrieval is done 10 minutes after the encoding, outside of the scanner. People are presented with the same 78 images in a new order and 39 new images, appearing one at a time in the center of the screen. They have to determine whether each image has been previously presented, and if 'Yes', where it was located.

OTHER OUTCOMES:
Transfer to everyday life (self-reported): Meta-memory rating | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  Mean scores from the Meta-memory questionnaire (MMQ).
Transfer to everyday life (self-reported): Attention and recent memory rating | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  Mean scores from the Auto-administered Memory Questionnaire (AMQ, short version).
Transfer to everyday life (self-reported): Activities of daily living | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  A composite score will be computed that aggregates the average z-scores from the participant + informant versions of the Alzheimer's Disease Cooperative Study - Activities of Daily Living - Prevention Instrument (ADCS-ADL-PI).
Transfer to everyday life (self-reported): Cognitive activities | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  Mean scores from the Cognitive Activities questionnaire.
Transfer to everyday life (self-reported): Jessen's Questions | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  The number of participants that do not have a memory complaint.
Transfer to everyday life (performance-based): Instrumental Activities of Daily Living | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  Mean scores from the Direct Assessment of Functional Status - Revised (DAFS-R), an ecologically-valid task assessing everyday life situations.
Transfer to everyday life (performance-based): Memory Strategies | PRE (within 12 weeks before intervention starts) + POST-1 (within 8 weeks after the end of intervention) + POST-2 (2 years from PRE, +/- 3 months)
  Mean scores from the Memory Toolbox Test, a questionnaire assessing the knowledge of memory strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Belleville, PhD, Principal Investigator — Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Locations (2):
- Canada (2):
  - Rotman Research Institute, Baycrest, Toronto, Ontario
  - CRIUGM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belleville S, Moussard A, Ansaldo AI, Belchior P, Bherer L, Bier N, Bohbot VD, Bruneau MA, Cuddy LL, Gilbert B, Jokel R, Mahalingam K, McGilton K, Murphy KJ, Naglie G, Rochon E, Troyer AK, Anderson ND. Rationale and protocol of the ENGAGE study: a double-blind randomized controlled preference trial using a comprehensive cohort design to measure the effect of a cognitive and leisure-based intervention in older adults with a memory complaint. Trials. 2019 May 22;20(1):282. doi: 10.1186/s13063-019-3250-6. PMID 31118095